CLINICAL TRIAL: NCT06705127
Title: A Phase II,Single-arm,Multicenter Study of Radiotherapy Followed by Chemotherapy Combined With Toripalimab Immunotherapy in Local Advanced HR-positive,HER2-negative Breast Cancer.
Brief Title: Radiotherapy Followed by Chemotherapy Combined With Toripalimab in Local Advanced HR-positive,HER2-negative BC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-114
Record Dates: First submitted 2024-11-24; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: HR-positive,HER2-negative Breast Cancer
Keywords: HR-positive,HER2-negative Breast Cancer; Local Advanced; Toripalimab; Radiotherapy; Neoadjuvant
MeSH Terms: interventions — Epirubicin; Cyclophosphamide; 130-nm albumin-bound paclitaxel; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab treatment group (Experimental): Local radiotherapy: Subjects received stereotactic radiotherapy for the primary breast cancer lesion at 8Gy each time for 3 consecutive days, once a day, 2 weeks before the start of systemic therapy.
  Drug A: 240mg intravenous infusion of Toripalimab, once every 3 weeks, the first dosing date was C1D1,followed by the first day of each course for 18 cycles, a total of 1 year.
  Drugs B and C: Epirubicin was administered intravenously after the dosage was calculated at 90mg/m2 body surface area, cyclophosphamide was calculated at 600mg/m2 body surface area by intravenous micropump, both drugs were administered every 3 weeks, the first administration date was C1D1, and then the first day of each course was administered for 4 cycles.
  Drug D: albumin paclitaxel was given intravenatically at a dose of 125mg/m2 body surface area, once a week, with the first administration date of C5D1, and then on the first day of each course for 12 cycles.
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 ); Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) — Drug A: 240mg intravenous infusion of Toripalimab, once every 3 weeks, the first dosing date was C1D1, followed by the first day of each course for 18 cycles, a total of 1 year.
  Drugs B and C: Epirubicin was administered intravenously after the dosage was calculated at 90mg/m2 body surface area, cyclophosphamide was calculated at 600mg/m2 body surface area by intravenous micropump, both drugs were administered every 3 weeks, the first administration date was C1D1, and then the first day of each course was administered for 4 cycles.
  Drug D:albumin paclitaxel was given intravenatically at a dose of 125mg/m2 body surface area, once a week, with the first administration date of C5D1, and then on the first day of each course for 12 cycles.
  Other Names: Epirubicin; cyclophosphamide; nab-paclitaxel
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Local radiotherapy: Subjects received stereotactic radiotherapy for the primary breast cancer lesion at 8Gy each time for 3 consecutive days, once a day, 2 weeks before the start of systemic therapy

SUMMARY:
This study is the first to explore the clinical study of neoadjuvant radiotherapy followed by chemotherapy combined with terriplizumab in breast cancer. Participants with locally advanced (T1c-T2(≥2cm) N1-2M0 or T3-4cN0-2M0) HR-positive and HER2-negative breast cancer were enrolled to evaluate the efficacy and safety of neoadjuvant radiotherapy followed by chemotherapy combined with triplimab in the treatment of locally advanced HR-positive and HER2-negative breast cancer. About 30 participants are planned to participate in this clinical study.

DETAILED DESCRIPTION:
Breast cancer is the first malignant tumor in women worldwide, and its incidence is still increasing year by year. Compared with developed countries in Europe and the United States, although the incidence of breast cancer in China is low, it is showing a rapid growth trend, and due to practical factors such as large population base and unbalanced distribution of medical resources, the overall stage of initial diagnosis of breast cancer patients in China is later than that in developed countries in Europe and the United States, and the proportion of local advanced and advanced breast cancer patients is higher. As the overall prognosis of early breast cancer patients is good, how to further improve the therapeutic effect of locally advanced and advanced breast cancer patients has become the main pass to improve the overall prognosis of breast cancer. In the comprehensive treatment strategy of breast cancer, radiotherapy is an indispensable part of local treatment. In the past, the understanding of the antitumor effect of radiotherapy was mainly limited to the dormancy or lytic death of tumor cells caused by DNA damage in tumor cells caused by X-ray. However, in recent years, with the deepening of research on tumor microenvironment and immunotherapy, researchers have gradually revealed the remodeling effect of radiotherapy on tumor microenvironment. We designed this clinical study of neoadjuvant radiotherapy sequential chemotherapy combined with terriplizumab immunotherapy to explore the effect of neoadjuvant radiotherapy sequential chemotherapy combined with terriplizumab on postoperative pCR rate and prognosis of patients with locally advanced HR-positive and HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Histologically or pathologically confirmed non-specific invasive ductal carcinoma, histologically grade3, ER≥1%, HER2 negative, Ki-67>20%;
3. T1c-T2(≥2cm)N1-2M0 or T3-4cN0-2M0;
4. No previous treatment;
5. ECOG PS 0-1 score;
6. The subject or legal representative has been informed of the nature of the study, understands the protocol, is able to guarantee compliance, and signs the informed consent

Exclusion Criteria:

1. Those who are known to be allergic to recombinant humanized antiPD-1 monoclonal antibody drugs and their components;
2. Currently participating in and receiving other research treatment;
3. Previously received systematic treatment for breast cancer, including systematic chemotherapy, targeted therapy, immunotherapy, etc.;
4. Remote metastatic lesions of breast cancer were confirmed by imaging or pathology;
5. Patients with active tuberculosis (TB) who are receiving anti-TB therapy or have received anti-TB therapy within 1 year prior to screening;
6. Uncontrolled or symptomatic hypercalcemia (> 1.5mmol/L calcium ion or calcium > 12mg/dL or corrected serum > ULN);
7. Clinically uncontrolled active infections, including but not limited to acute pneumonia;
8. Uncontrollable major seizures or superior vena cava syndrome;
9. previous or current co-occurrence of other malignant tumors (except for non-melanoma skin basal cell carcinoma or squamous cell carcinoma, breast/cervical carcinoma in situ, superficial bladder carcinoma and other in situ cancers that have been treated radically and have no evidence of disease recurrence);
10. Have a history of interstitial pneumonia, idiopathic pulmonary fibrosis, institutional pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, chest CT screening found evidence of active pneumonia or other moderate to severe lung diseases that seriously affect lung function;
11. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive);
12. Severe cardiovascular disease, such as New York Heart Association (NYHA) grade 2 or higher heart failure, unstable angina, unstable arrhythmia, myocardial infarction or cerebrovascular accident within the first 6 months of enrollment;
13. received systemic immunosuppressive drugs (i.e. use of corticosteroids or immunosuppressive drugs) for any active autoimmune disease within 2 years prior to study initiation;
14. Received live virus vaccine within 4 weeks prior to study initiation;
15. Patients who have previously received allogeneic stem cells or parenchymal organ transplants;
16. Pregnant or lactating women or women who have the possibility of becoming pregnant have tested positive for pregnancy before the first drug use, and patients who are fertile but do not want to take contraceptive measures or their sexual partners do not want to take contraceptive measures
17. Any other clinically significant illness or condition that the investigator believes could affect adherence to the protocol (such as a history of mental illness or substance abuse), prevent the patient from benefiting from the clinical study, or prevent the patient from signing informed consent (such as drug use and substance abuse), or make participation in the clinical study inappropriate (including but not limited to: Abnormal laboratory results, clinical active diverticulitis, abdominal abscess, intestinal obstruction, and peritoneal metastases).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response（pCR） | Up to12 months
  pCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peifen Fu, MD, Principal Investigator — Zhejiang University; Senxiang Yan, MD, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No